CLINICAL TRIAL: NCT05552859
Title: A 24-Week, Multicenter, Randomized, Open-Label, Parallel-Group Trial Comparing the Efficacy and Safety of Insulin Glargine 300 U/mL (Gla-300) and Insulin Degludec 100 U/mL (IDeg-100) in Insulin-Naïve People With Type 2 Diabetes Mellitus and Renal Impairment: TRENT Trial
Brief Title: Gla-300 and IDeg-100 in Insulin-Naïve People With Type 2 Diabetes Mellitus and Renal Impairment
Acronym: TRENT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision to cancel trial due to poor recruitment/ severe recruitment delay and not related to safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS17007; 2022-001485-35 (EudraCT Number)
Record Dates: First submitted 2022-09-07; First posted 2022-09-23 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus; Renal Impairment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — Insulin Glargine; insulin degludec

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gla-300 arm (Experimental): Gla-300 will be administered once daily for 24 weeks
  Interventions: Drug: Insulin glargine 300 U/mL
- IDeg-100 arm (Active Comparator): Ideg-100 will be administered once daily for 24 weeks
  Interventions: Drug: Insulin degludec 100 U/mL

INTERVENTIONS:
Drug: Insulin glargine 300 U/mL — Insulin glargine 300 U/mL in the SoloStar pen, self-administered once daily for 24 weeks.
  Other Names: Toujeo; HOE901-U300
  Arms: Gla-300 arm
Drug: Insulin degludec 100 U/mL — Insulin degludec 100 U/mL will be self- administered once daily for 24 weeks.
  Other Names: Tresiba
  Arms: IDeg-100 arm

SUMMARY:
The TRENT trial is designed to confirm the efficacy and safety of Gla-300 compared with IDeg-100 in insulin-naïve patient (participants who have not tried insulin) with Type 2 Diabetes Mellitus (T2DM) and renal impairment. It will test the hypothesis that Gla-300 is non-inferior to IDeg-100 with glucose control. If achieved, the trial will also test for the superiority of Gla-300 compared with IDeg-100 in Hemoglobin A1c (HbA1c) reduction, without an increased potential risk of hypoglycemia.

DETAILED DESCRIPTION:
The trial will consist of the following periods:

* A screening period of up to 2 weeks,
* A 24-week, open-label treatment period, including a titration period and a maintenance period.
* A 7-day, post-treatment, safety follow-up period after the last dose of the study drug or after premature/permanent discontinuation from study drug treatment. This will be a phone contact, but could be a site visit if ongoing or new AEs emerge during the post-treatment period, if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Is an adult aged ≥18 years at screening.
2. Was diagnosed with Type 2 Diabetes Mellitus (T2DM) of >1-year duration and had glycemic levels above target with OADs (Oral Antidiabetic Drug) with or without GLP-1 RA (glucagon-like peptide-1 receptor agonist) (oral or injectable) at stable doses for ≥3 months before the screening period.
3. Has an HbA1c ≥7.5% and ≤10.5% at screening.
4. Has renal impairment, as defined by an eGFR (estimated glomerular filtration rate) of <60 mL/min/1.73m2 and ≥15 mL/min/1.73m2.
5. Has adequately controlled blood pressure with stable antihypertensive therapy at trial inclusion.
6. Is insulin-naïve, except for short use of insulin not exceeding 15 days during the last year before the screening period.
7. Is capable of understanding the written informed consent, and provides signed written informed consent.
8. Is willing and able to complete the electronic diary (eDiary) and agrees to comply with protocol requirements.
9. Is willing and able to fast without having administered study drug for scheduled site visits.

Exclusion Criteria:

1. Has initiated treatment with potential novel therapies like dual glucose-dependent insulinotropic polypeptide (GIP) and GLP-1 RA.
2. Has a body mass index (BMI)* >45 kg/m² during the screening period.
3. Has a history of hypoglycemia unawareness (defined as the onset of neuroglycopenia before the appearance of autonomic warning symptoms [eg, blurred vision, difficulty speaking, feeling faint, difficulty thinking, and confusion] or as the failure to sense a significant fall in blood glucose below normal levels).
4. Has a history of 2 or more episodes of severe hypoglycemia and/or 2 or more episodes of diabetic ketoacidosis within the 6 months before the day of screening.
5. Has been exposed to other investigational drug(s) within 1 month or 5 half-lives from screening, whichever is longer.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-08-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (68):
- United States (32):
  - Yuma Clinical Trials, LLC Site Number: 8400028, Yuma, Arizona
  - American Clinical Trials Site Number: 8400014, Buena Park, California
  - Clearview Medical Research LLC Site Number: 8400021, Canyon Country, California
  - Torrance Clinical Research Institute Site Number: 8400003, Lomita, California
  - Center for Endocrinology Diabetes and Metabolic Disorders (CEDMD) - CAR Site Number: 8400026, Santa Clarita, California
  - San Fernando Valley Health Institute - ClinEdge - PPDS Site Number: 8400023, Van Nuys, California
  - Chase Medical Research LLC Site Number: 8400007, Waterbury, Connecticut
  - Innovative Research of West Florida Site Number: 8400016, Clearwater, Florida
  - Evolution Clinical Trials Site number: 8400034, Hialeah Gardens, Florida
  - Wellness Research Center Inc - Miami Site Number: 8400010, Miami, Florida
  - Med Research of Florida, LLC Investigator Site: 8400033, Miami, Florida
  - Florida Institute For Clinical Research LLC Site Number: 8400004, Orlando, Florida
  - Emory University Site Number: 8400032, Atlanta, Georgia
  - Agile Clinical Research Trials, LLC Site Number: 8400001, Atlanta, Georgia
  - Centricity Research Site Number: 8400006, Columbus, Georgia
  - Georgia Clinical Research Site Number: 8400009, Lawrenceville, Georgia
  - Endocrine and Metabolic Consultants Research Center Site Number: 8400031, Rockville, Maryland
  - Diabetes, Obesity, Cardiovascular Clinical Specialists (DOCS) Site Number: 8400019, Las Vegas, Nevada
  - Mid Hudson Medical Research PLLC Site Number: 8400024, New Windsor, New York
  - Lucas Research - Morehead City - HyperCore - PPDS Site Number: 8400008, Morehead City, North Carolina
  - Advanced Medical Research Site Number: 8400012, Maumee, Ohio
  - Capital Area Research LLC Site Number: 8400029, Newport, Pennsylvania
  - Jefferson University Physicians (JUP) Site Number: 8400025, Philadelphia, Pennsylvania
  - Holston Medical Group PC Site Number: 8400018, Bristol, Tennessee
  - Frontier Medical Center Site Number: 8400035, El Paso, Texas
  - Diabetes and Thyroid Center of Fort Worth PLLC Site Number: 8400015, Fort Worth, Texas
  - Juno Research, LLC Site Number: 8400017, Houston, Texas
  - Reichman and Associates Site Number: 8400013, Houston, Texas
  - Texas Institute for Kidney and Endocrine Disorders Site Number: 8400027, Lufkin, Texas
  - Northeast Clinical Research of San Antonio LLC Site Number: 8400022, Schertz, Texas
  - Consano Clinical Research Site Number: 8400030, Shavano Park, Texas
  - David Ramstad Associates Research - IACT - HyperCore - PPDS Site Number: 8400005, Suffolk, Virginia
- Czechia (6):
  - Diabetologie MUDr. Tomas Edelsberger Site Number: 2030001, Krnov, Moravskoslezský kraj
  - Agentura Science Pro spol. s.r.o.Site Number: 2030002, Olomouc, Olomoucký kraj
  - Institut Klinicke A Experimentalni Mediciny Site Number: 2030006, Prague, Praha, Hlavní Mesto
  - Diacentrum Brandys n. L. Site Number: 2030004, Brandýs nad Labem-Stará Boleslav
  - Diabetologicka, interni a obezitologicka ambulance Site Number: 2030005, Jílové u Prahy
  - Fakultni nemocnice Kralovske Vinohrady Site Number: 2030007, Prague
- Hungary (6):
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz Site Number: 3480006, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Markusovszky Egyetemi Oktatókórház Site Number: 3480001, Szombathely, Vas County
  - Csolnoky Ferenc Korhaz Site Number: 3480005, Balatonfüred, Veszprém megye
  - Zala Megyei Szent Rafael Korhaz Site Number: 3480002, Zalaegerszeg, Zala County
  - Magyar Honvédség Egészségügyi Központ Site Number: 3480003, Budapest
  - Somogy Megyei Kaposi Mór Oktató Kórház Site Number: 3480004, Kaposvár
- Poland (18):
  - Centrum Medyczne OMEDICA Site Number: 6160013, Poznan, Greater Poland Voivodeship
  - Zaklad Opieki Medycznej "Sanatio" Sp.z o.o. - Osrodek Leczenia Schorzen Cywilizacyjnych Site Number: 6160016, Krakow, Lesser Poland Voivodeship
  - Regionalna Poradnia Diabetologiczna - Wroclaw Site Number: 6160009, Wroclaw, Lower Silesian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Przychodnia Specjalistyczna Medica Site Number: 6160008, Lublin, Lublin Voivodeship
  - KO-MED Centra Kliniczne Sp. z o.o. Site Number: 6160010, Puławy, Lublin Voivodeship
  - KO-MED Centra Kliniczne Sp. z o.o. Site Number: 6160012, Zamość, Lublin Voivodeship
  - Prywatny Gabinet Lekarski Centrum Medyczne Diabetika Dorota Mlodawska-Choluj Site Number: 6160015, Radom, Masovian Voivodeship
  - NBR Polska Site Number: 6160003, Warsaw, Masovian Voivodeship
  - Centralny Szpital Kliniczny MSW Site Number: 6160005, Warsaw, Masovian Voivodeship
  - NZOZ Gdanska Poradnia Cukrzycowa Sp. z o.o. Site Number: 6160014, Gdansk, Pomeranian Voivodeship
  - NZOZ Specjalistyczny Osrodek Internistyczno-Diabetologiczny Site Number: 6160001, Częstochowa, Silesian Voivodeship
  - Specjalistyczna Praktyka Lekarska Site Number: 6160004, Lubliniec, Silesian Voivodeship
  - ETG Lodz Site Number: 6160018, Lodz
  - Gabinet Lekarski Malgorzata Saryusz-Wolska Site Number: 6160017, Lódz
  - Praktyka Lekarska Ewa Krzyzagórska Site Number: 6160014, Poznan
  - Prywatny Gabinet Lekarski, Centrum Medyczne "Diabetika" Site Number:6160002, Radom
  - ETG Skierniewice - PPDS Site Number: 6160006, Skierniewice
  - KO-MED Centra Kliniczne Sp. z o.o. Site Number:6160011, Staszów, Świętokrzyskie Voivodeship
- Serbia (6):
  - Clinical Hospital Centar Zvezdara Site Number: 6880001, Belgrade
  - University Clinical Center of Serbia - PPDS Site Number: 6880003, Belgrade
  - University Clinical Center of Serbia - PPDS Site Number: 6880004, Belgrade
  - University Clinical Center Nis Site Number: 6880002, Niš
  - University Clinical Center Nis Site Number: 6880005, Niš
  - Health Center Zajecar Site Number: 6880006, Zaječar

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS17007 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25294&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 68 study centers across 5 countries. A total of 182 participants were screened between 05 December 2022 and 30 June 2023, of whom 120 were screen failures. The number of randomized participants remained significantly lower (<10%) than was originally planned. Consequently, the estimated results would have been delayed by several years. Hence, the sponsor made the strategic decision to discontinue the trial due to this significant recruitment delay, not related safety.
Pre-assignment Details: A total of 62 participants were randomized in 1:1 ratio to either Gla-300 group, or IDeg-100 group, stratified by screening glycated hemoglobin (HbA1c) values (<8.5% or ≥ 8.5%); and use of sulfonylurea (SU) before the day of screening ('yes' versus 'no').There were no safety signals detected, and the study team remained blinded to the data collected for the randomized subjects at the time of the study termination decision.
Groups:
- Gla-300 U/mL Arm: Gla-300 will be administered once daily for 24 weeks
  Insulin glargine 300 U/mL: Insulin glargine 300 U/mL in the SoloStar pen, self-administered once daily for 24 weeks.
- IDeg-100 U/mL Arm: Ideg-100 will be administered once daily for 24 weeks
  Insulin degludec 100 U/mL: Insulin degludec 100 U/mL will be self- administered once daily for 24 weeks.
Period: Overall Study
Arm/Group | Gla-300 U/mL Arm | IDeg-100 U/mL Arm
Started | 31 | 31
Completed (Sanofi LPS17007 study was terminated by the Sponsor due to poor recruitment/severe recruitment delay and was not related to safety concern.) | 1 | 1
Not Completed | 30 | 30
Not completed — Study was terminated by the Sponsor due to poor recruitment/severe recruitment delay | 30 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gla-300 Arm | IDeg-100 Arm | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (7.5) | 71.0 (7.7) | 71.5 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 29 | 25 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 27 | 29 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Hungary | 3 | 6 | 9
  United States | 7 | 9 | 16
  Czechia | 5 | 3 | 8
  Poland | 12 | 9 | 21
  Serbia | 4 | 4 | 8
Weight (kg) [Mean (Standard Deviation); unit: kg] | 89.5 (25.30) | 89.5 (20.32) | 89.5 (22.74)
BMI (kg//m²) [Mean (Standard Deviation); unit: (kg/m²)] | 31.6 (5.54) | 32.2 (6.56) | 31.9 (6.03)
BMI by category (kg/m²) [Count of Participants; unit: Participants] — Number of participants with a BMI <30 or ≥30 (kg/m2)
  Participants
    <30 | 13 | 15 | 28
    ≥30 | 18 | 16 | 34
Baseline HbA1c (%) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c: glycated hemoglobin
  Percentage of HbA1c | 8.4 (0.74) | 8.4 (0.72) | 8.4 (0.72)
Baseline HbA1c (%) group [Count of Participants; unit: Participants] — Number of Patients with <8.5 or ≥8.5 HbA1c (glycated hemoglobin).
  Participants
    <8.5 | 20 | 19 | 39
    ≥8.5 | 11 | 12 | 23
Baseline FPG (mg/dL) [Mean (Standard Deviation); unit: (mg/dL)] — FPG: fasting plasma glucose Population: Baseline FPG was missing 2 participants (1 participant in the Gla-300 and 1 in the IDeg-100 Arm).
  (mg/dL)
    number analyzed (Participants) | 30 | 30 | 60
    (all) | 162.8 (28.14) | 170.5 (36.20) | 166.7 (32.38)
Baseline SMPG (mg/dL) [Mean (Standard Deviation); unit: (mg/dL)] — SMPG: self-measured plasma glucose Population: Baseline SMPG was missing from 13 participants (Gla-300 Arm) and from 20 participants (IDeg-100 arm).
  (mg/dL)
    number analyzed (Participants) | 18 | 11 | 29
    (all) | 153.9 (30.45) | 169.0 (50.03) | 159.6 (38.90)
eGFR (mL/min/1.73m²) [Mean (Standard Deviation); unit: (mL/min/1.73m²)] — eGFR: estimated glomerular filtration rate.
  (mL/min/1.73m²) | 45.7 (9.6) | 47.8 (11.2) | 46.7 (10.4)
eGFR (mL/min/1.73m²) [Count of Participants; unit: Participants] — Number of participants with eGFR of <45 or ≥45.
  Participants
    <45 | 13 | 11 | 24
    ≥45 | 18 | 20 | 38
Antihyperglycemic therapies [Count of Participants; unit: Participants] — Percentages were based on n or N.
  Participants
    SU (sulfonylurea) | 17 | 15 | 32
    Metformin | 22 | 21 | 43
    GLP-1 RA (glucagon-like peptide-1 receptor agonist) | 5 | 2 | 7
    Dipeptidyl peptidase IV inhibitors/gliptin | 6 | 6 | 12
    SGLT-2i (sodium-glucose co-transporter-2 inhibitors) use | 16 | 12 | 28
    Thiazolidinediones/glitazones | 2 | 5 | 7
Age (years) at diagnosis of diabetes [Mean (Standard Deviation); unit: years] | 59.0 (9.2) | 55.9 (8.2) | 57.5 (8.8)
Duration of diabetes (time since diagnosis) (years) [Mean (Standard Deviation); unit: years] | 13.6 (7.2) | 15.6 (8.3) | 14.6 (7.8)
History of gestational diabetes [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 0
  No | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Mean Change From Baseline to Week 24 in HbA1c Level (Gla-300 vs IDeg-100)
Description: Change in HbA1c was calculated by subtracting baseline value from Week 24 value and then mean values were calculated.
Time Frame: Baseline to 24 weeks
Population: In the Gla-300 arm, 8 participants were in the predefined Analysis Window for the 24 weeks assessment. In the IDeg-100 Arm, 9 participants were within the predefined Analysis Window for the 24 weeks assessment. These 8 and 9 participants did not complete the 24 weeks treatment period.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Gla-300 U/mL Arm | IDeg-100 U/mL Arm
Number analyzed (Participants) | 8 | 9
percentage of HbA1c | -0.4 (1.73) | -1.0 (0.98)

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 24
Description: Change in FPG was calculated by subtracting baseline value from the Week 24 value.
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: (mg/dL)
Arm/Group | Gla-300 U/mL Arm | IDeg-100 U/mL Arm
Number analyzed (Participants) | 7 | 9
(mg/dL) | -36.4 (25.16) | -55.5 (22.67)

3. Secondary Outcome: Change in Fasting Self-Measured Plasma Glucose (SMPG) From Baseline to Week 24
Description: Change in SMPG was calculated by subtracting baseline value from the Week 24 value.
Time Frame: Baseline to 24 weeks
Population: Due to early trial termination, a meaningful comparison of the mean (SD) change in fasting SMPG (expressed in both mg/dL and mmol/L) was not possible because of the small sample size in both treatment groups, especially at Week 24.
Measure: Mean (Standard Deviation); unit: (mmol/L)
Arm/Group | Gla-300 U/mL Arm | IDeg-100 U/mL Arm
Number analyzed (Participants) | 1 | 0
(mmol/L) | -4.00 |

4. Secondary Outcome: Change in 7-point SMPG Profiles From Baseline to Week 24, Per Time Point Within 24-hour Period
Description: 7-point SMPG profiles were measured at the following 7 points: pre-breakfast, 2 hours after breakfast, pre-lunch, 2 hours after lunch, pre-dinner, 2 hours after dinner, and bedtime.
Time Frame: Baseline to 24 weeks
Population: Due to early trial termination, a meaningful comparison of the mean (SD) change in 7-point SMPG profile (expressed in both mg/dL and mmol/L) at 7 time points within a 24-hour period was not possible because of the small sample size in both treatment groups, especially at Week 24.
Measure: Mean (Standard Deviation); unit: (mmol/L)
Arm/Group | Gla-300 U/mL Arm | IDeg-100 U/mL Arm
Number analyzed (Participants) | 1 | 0
(mmol/L)
  7-Point SMPG Profile (mmol/L), before breakfast (fasting) | -4.13 |
  7-Point SMPG Profile (mmol/L), 2 hours after breakfast | -1.30 |
  7-Point SMPG Profile (mmol/L), before lunch | 0.31 |
  7-Point SMPG Profile (mmol/L), 2 hours after lunch | 0.63 |
  7-Point SMPG Profile (mmol/L), before dinner | 2.18 |
  7-Point SMPG Profile (mmol/L), 2 hours after dinner | -5.36 |
  7-Point SMPG Profile (mmol/L), at bedtime | -6.20 |

5. Secondary Outcome: Percentage of Participants Reaching HbA1c Target of <7.0% at Week 24
Description: If a patient has a missing HbA1c value at Week 24, it is assumed that they did not reach the HbA1c target of <7.0%.
  HbA1c value of 7.0% is equivalent to 53.0 mmol/mol.
Time Frame: At week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Gla-300 U/mL Arm | IDeg-100 U/mL Arm
Number analyzed (Participants) | 31 | 31
Participants | 4 | 2

6. Secondary Outcome: Percentage of Participants With ≥1 Episode(s) of Confirmed Hypoglycemia Event (Cut-off Value 70 mg/dL and 54 mg/dL) During the 24-week Treatment Period.
Description: Any event recorded with Yes as response to the question, "Was a glucose measurement obtained at the time of the event before countermeasure?" and a measurable glucose level of <70 mg/dL. ADA (American Diabetes Association), Level 1 was defined as a measurable glucose concentration of <70 mg/dL (3.9 mmol/L) but ≥54 mg/dL (3.0 mmol/L).
Time Frame: Baseline to end of study (25 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Gla-300 U/mL Arm | IDeg-100 U/mL Arm
Number analyzed (Participants) | 11 | 9
percentage of participants | 35.5 | 29.0

7. Secondary Outcome: Rate of Hypoglycemia Per Participant-year
Description: Computed as: 365.25/12 × (number of episodes of hypoglycemia)/(number of days exposed in time window)
Time Frame: Baseline to end of study (25 weeks)]
Measure: Number; unit: Rate of hypoglycemia per patient-year
Arm/Group | Gla-300 U/mL Arm | IDeg-100 U/mL Arm
Number analyzed (Participants) | 31 | 31
Rate of hypoglycemia per patient-year | 9.5 | 5.6

8. Secondary Outcome: Percentage of Participants and Event Rate of Hypoglycemia by Trial Period (for ≤12 Weeks, for >13 Weeks to ≤24 Weeks)
Description: Hypoglycemic events measured at the following intervals: Weeks 1-12 and Weeks 13-24.
Time Frame: Baseline to end of study (25 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Gla-300 U/mL Arm | IDeg-100 U/mL Arm
Number analyzed (Participants) | 31 | 31
Participants
  Titration period (Week 1 to Week 12) | 9 | 7
  Maintenance period (Week 13 to Week 24) | 5 | 5

9. Secondary Outcome: The 24-hour (All Time), Occurrence of Each Episode of Documented Hypoglycemia by Category, Presented by 2-hour Timeframe Over 24 Hours During the 24-week Treatment Period.
Description: The time range for this outcome measure was 00:00 to 05:59, both inclusive. Hypoglycemia Categories [(symptomatic, asymptomatic, severe) are defined per the American Diabetes Association/European Association for the Study of Diabetes hypoglycemia Classification]
Time Frame: Baseline to end of study (25 weeks)
Measure: Number; unit: Episodes
Arm/Group | Gla-300 U/mL Arm | IDeg-100 U/mL Arm
Number analyzed (Participants) | 31 | 31
Episodes | 11 | 9

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)) and Serious Adverse Events (SAEs), Including Adverse Events of Special Interest (AESIs)
Description: Adverse events (AEs) and serious adverse events (SAEs), including adverse events of special interest (AESIs), and other safety evaluations, including vital signs and body weight.
Time Frame: Baseline to end of study (25 weeks)
Population: Overall, 5 participants (16.1%) in the Gla-300 group reported 6 events, and 7 participants (22.6%) in the IDeg-100 group 16 events during the trial period. Note: in the Ideg group, 2 participants had both an AE and SAE.
Measure: Count of Participants; unit: Participants
Arm/Group | Gla-300 U/mL Arm | IDeg-100 U/mL Arm
Number analyzed (Participants) | 31 | 31
Participants
  Adverse Event (AE) | 5 | 7
  Serious Adverse Event | 1 | 3
  Adverse Event of Special Interest (AESIs) | 0 | 0
  Treatment-Emergent SAEs | 1 | 3

ADVERSE EVENTS:
Time Frame: All AEs (serious or nonserious) will be recorded from the signing of the ICF until the safety follow-up visit, patient's permanent discontinuation from the trial, or loss to follow-up, up to 25 weeks.
Arm/Group | Gla-300 U/mL Arm | IDeg-100 U/mL Arm
All-Cause Mortality (participants affected / at risk) | 0/31 | 1/31
Serious Adverse Events (participants affected / at risk) | 1/31 | 3/31
Other Adverse Events (participants affected / at risk) | 0/31 | 5/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gla-300 U/mL Arm (N=31) | IDeg-100 U/mL Arm (N=31)
Hypertensive Heart Disease (Cardiac disorders) | 0 (0) | 1 (1)
Hypoglycemic Event (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gla-300 U/mL Arm (N=31) | IDeg-100 U/mL Arm (N=31)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
The sponsor made the strategic decision to discontinue the trial due to a significant recruitment delay (ie, the number of randomized participants remained significantly lower [<10% than originally planned sample size]). No safety signals were detected during the trial, and the trial team remained blinded to the data collected for the randomized participants at the time of early discontinuation of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT05552859/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT05552859/SAP_001.pdf